CLINICAL TRIAL: NCT05277779
Title: EARLY Assessment of MYOcardial Tissue Characteristics in OBESITY (EARLY-MYO-OBESITY)
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Ningbo Hangzhou Bay Hospital (Unknown); Shanghai Jiading Central Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: ACFO2021
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2022-02

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control: non-obese （BMI<25kg/m2）controls without known endocrine diseases, cardiac disease, or other comorbidities, and with unremarkable imaging results.
  Interventions: Diagnostic Test: cardiac magnetic resonance(CMR)
- metabolically healthy obese: obese individuals having no more than one of the metabolic syndrome components (with exception of increased waist circumference) and without impaired glucose tolerance (defined as a 2-hour post loading glucose level of 7.7-11.1mmol/L )
  Interventions: Diagnostic Test: cardiac magnetic resonance(CMR)
- metabolically unhealthy obese: obese individuals with more than one metabolic syndrome components or impaired glucose tolerance
  Interventions: Diagnostic Test: cardiac magnetic resonance(CMR)

INTERVENTIONS:
Diagnostic Test: cardiac magnetic resonance(CMR) — CMR was performed to assess myocardial tissue characteristics in the study population

SUMMARY:
EARLY-MYO-OBESITY-CMR is a prospective, three-center, cardiac imaging study to investigate cardiac morphology, function, and tissue phenotypes in a cohort of non-diabetic obese adults, and compare with metabolically healthy non-obese controls.

DETAILED DESCRIPTION:
1. Transthoracic echocardiography was performed to analyze the LV morphology and function.
2. CMR was performed within 24 hours of the echocardiographic examination to assess the cardiac morphology , cardiac function, and myocardial tissue characteristics. Standard cine images were acquired to quantify LV function and volume. T1 mapping-derived ECV values were used to detect subtle diffuse fibrosis , and late gadolinium-enhanced (LGE) imaging was used to identify focal fibrosis. Native T2 values were obtained to quantify myocardial edema . Global longitudinal peak systolic strain (GLS) and e' SR were assessed by tissue tracking analysis to detect subclinical systolic and diastolic dysfunction.

ELIGIBILITY:
Inclusion criteria:

* age 18-75 years without cardiac symptoms or known cardiac diseas;
* body mass index ≥25 kg/m2

Exclusion criteria:

* coronary artery disease (coronary artery stenosis >50% on angiography or coronary computed tomography, documented myocardial infarction, or a history of coronary artery bypass graft surgery or percutaneous coronary intervention)
* non-ischemic cardiovascular disease, such as idiopathic cardiomyopathy, valvular disease, congenital heart disease, or pulmonary heart diseas
* a left ventricular (LV) ejection fraction of<50% on echocardiography or a history of heart failure
* arrhythmia or the presence of bundle branch block on electrocardiography
* pacemaker or defibrillator implantation
* renal dysfunction with an estimated glomerular filtration rate of <60 mL/min/1.73 m2
* contraindications to cardiac magnetic resonance (CMR) imaging
* malignancy or life expectancy of less than 2 year
* inability to provide written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult obese participants without cardiac symptoms or known cardiac disease
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
investigate cardiac morphology and function by CMR | 24 hours within recruitment
  cardiac morphology and function were assessed by CMR steady-state free precession sequences
investigate cardiac tissue characteristics by CMR | 24 hours within recruitment
  myocardial edema and fibrosis were assessed by CMR T2 mapping and ECV

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, Study Director — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao H, Huang R, Jiang M, Wang W, Chai Y, Liu Q, Zhang W, Han Y, Yan F, Lu Q, Tao Z, Wu Q, Yue J, Ma J, Pu J. Myocardial Tissue-Level Characteristics of Adults With Metabolically Healthy Obesity. JACC Cardiovasc Imaging. 2023 Jul;16(7):889-901. doi: 10.1016/j.jcmg.2023.01.022. Epub 2023 Apr 12. PMID 37052557